CLINICAL TRIAL: NCT00346762
Title: Host and Viral Factors in HIV-1-Infected Typical Progressors and Long-Term Survivors Among Former Blood Donors in Anhui Province, China
Brief Title: Evaluating Host and Viral Factors Among HIV Infected Former Commercial Blood Donors in Fuyang, Anhui Province, China
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Comprehensive International Program of Research on AIDS (Other)
Responsible Party: Sponsor
Other Study IDs: CIPRA CH 003; CIPRA; Project 3; 10402 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2006-06-29; First posted 2006-06-30 (Estimated); Last update posted 2014-05-19 (Estimated); Status verified 2014-05

CONDITIONS: HIV Infections
Keywords: Former Plasma Donors; Commercial Plasma Donors; Long-Term Nonprogressors; Host Factors; Viral Factors; HIV
MeSH Terms: conditions — HIV Infections | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood and urine

GROUPS / COHORTS (1):
- 1: HIV infected former commercial blood donors (FBDs) in Fuyang, Anhui Province
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — HIV prevention education and risk reduction counselig

SUMMARY:
HIV infected former commercial blood donors (FBDs) in Fuyang, Anhui Province, China were infected with HIV from a common-source exposure to contaminated blood. The purpose of this study is to examine the role of host and viral factors in HIV disease progression in this unique HIV infected population.

DETAILED DESCRIPTION:
The HIV epidemic in China has reached a phase of exponential growth. Among the infected are FBDs in rural communities, who became infected through contaminated blood collection equipment. In Fuyang, Anhui Province, China, unregulated commercial blood collection occurred from 1992 to 1995; during the last decade or so, some HIV infected FBDs have progressed to AIDS, while others are long-term nonprogressors, not requiring antiretroviral therapy (ART). Since the HIV infected participants in this study are predicted to have been infected by the same or related HIV strain because of their location and how they were infected, this is a unique population to study. It is hypothesized that host factors, such as host immunity and genetic background, are better predictors of disease progression than viral factors in this population. This study will enroll HIV-1 infected FBDs and age-matched HIV uninfected adults in Fuyang, Anhui Province, China.

There are two stages in this study. Stage I is a cross-sectional study and will last 3 months. Participants will be HIV-1 infected FBDs and age-matched HIV uninfected controls. There are two study visits in Stage I; there will be a 2-day screening/enrollment visit and a follow-up visit. On the first day of screening/enrollment, participants will be briefed about the study and will be asked to complete demographic and risk factor questionnaires; medical and medication history will be reviewed and a physical examination will also occur. All participants will receive HIV prevention education and risk reduction counseling; additionally, HIV uninfected participants will receive HIV pretest counseling. On the second day of screening, participants will return to the clinic for blood collection, and females will undergo a pregnancy test. All participants will return to the clinic to receive their laboratory results and post-test counseling at a follow-up visit occurring approximately 2 weeks after their screening/enrollment visit. Any participant with a CD4 count less than 200 cells/mm3 or meeting other China Comprehensive AIDS Response (CARES) treatment criteria will be referred for further evaluation and care. HIV infected FBD participants with a CD4 count of 200 cells/mm3 or more will be invited to enroll in Stage II.

Stage II is a longitudinal, prospective study and will last 19.5 months. Stage II will enroll eligible HIV infected participants from Stage I and if necessary, other eligible patients referred from China CARES. There will be at least five study visits; they will occur at a 2-day study screening/enrollment visit, a follow-up visit 2 weeks after screening/enrollment, and Months 6, 12, and 18. Screening/enrollment and follow-up visit procedures will be identical to those conducted in Stage I. Visits at Months 6, 12, and 18 will occur over 2-day periods. Medical and medication history will be reviewed and a physical examination will occur on the first day; participants will need to return to the clinic for blood collection on the second day. Participants will receive laboratory results and post-test counseling at the next scheduled study visit. Additional study visits may be required if a participant experiences any clinically significant condition during the study.

ELIGIBILITY:
Inclusion Criteria for Stage I HIV Infected FBDs:

* Self-reported history of blood donation in 1995 or before
* HIV-1 infected
* ART naive
* Willing to provide locator information
* Willing to use acceptable forms of contraception

Inclusion Criteria for Stage I HIV Uninfected Controls:

* HIV uninfected
* Willing to provide locator information
* Willing to undergo repeat HIV testing

Inclusion Criteria for Stage II:

* Participant of Stage I OR enrolled directly from the ongoing China CARES program
* Self-reported history of blood donation in 1995 or before
* HIV-1 infected
* CD4 count of 200 cells/mm³ or more
* ART naive and willing to notify study staff prior to initiating any ART
* Clinical Stage I or II by the World Health Organization (WHO) Staging System
* Willing to adhere to the study follow-up schedule
* Willing to provide locator information
* Willing to use acceptable forms of contraception

Exclusion Criteria for All Participants:

* Concomitant use of ART during the study
* Pregnancy

Exclusion Criteria for Stage II:

* Plan to leave study area for more than 6 months during the follow-up period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample of HIV infected and uninfected blood donors
Sampling Method: Non-Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2005-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Change in CD4 count | At Month 3
Progression of HIV-1 disease | At Month 22

CONTACTS AND LOCATIONS:
Overall Officials: Yiming Shao, MD, PhD, Study Chair — National Center for AIDS/STD Control and Prevention (NCAIDS), Chinese Center for Disease Control and Prevention (China CDC); Jianqing Xu, MD, PhD, Principal Investigator — National Center for AIDS/STD Control and Prevention (NCAIDS), Chinese Center for Disease Control and Prevention (China CDC); Hui Xing, MD, MS, Principal Investigator — National Center for AIDS/STD Control and Prevention (NCAIDS), Chinese Center for Disease Control and Prevention (China CDC); Yuhua Ruan, PhD, Principal Investigator — National Center for AIDS/STD Control and Prevention (NCAIDS), Chinese Center for Disease Control and Prevention (China CDC); Jianjun Wang, MPH, Principal Investigator — Anhui Provincial Center for Disease Control and Prevention
Locations (1):
- Fuyang Prefecture Endemic Station, Anhui Province CIPRA CRS, Beijing, China

REFERENCES:
- [Background] Wu Z, Rou K, Cui H. The HIV/AIDS epidemic in China: history, current strategies and future challenges. AIDS Educ Prev. 2004 Jun;16(3 Suppl A):7-17. doi: 10.1521/aeap.16.3.5.7.35521. PMID 15262561
- [Result] Xu JQ, Wang JJ, Han LF, Xu C, Ruan YH, Xu ZH, Chen X, Liu ZD, Wang J, Su B, Ding XP, Gao B, Gu YB, Cao XY, Xing H, Hong KX, Peng H, Zhao QB, Yuan L, Feng Y, Zhang GY, Ma LY, Wu L, Shao YM. Epidemiology, clinical and laboratory characteristics of currently alive HIV-1 infected former blood donors naive to antiretroviral therapy in Anhui Province, China. Chin Med J (Engl). 2006 Dec 5;119(23):1941-8. PMID 17199937